CLINICAL TRIAL: NCT05226676
Title: Long-term Effects of Repetitive TMS in Chronic Neuropathic Pain in People With SCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI left the institution and the study couldn't be transfer to a new PI
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Maria Del Mar Cortes, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-20-00230; 19-1382-00001-01-PD (Other Grant/Funding Number: New York State Department Of Health)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries; Neuralgia; Chronic Pain
Keywords: Spinal Cord Injuries; Neuropathic; Chronic Pain; Transcranial Magnetic Stimulation; Neural Plasticity; Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Chronic Pain; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized double blinded sham controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real rTMS group (Experimental): Repetitive TMS at 20Hz frequency over the M1 will be performed for five consecutive days for 2 weeks (using 90% of the resting motor threshold/total of 500 pulses). The rTMS will be applied through a figure-8 coil connected to a magnetic stimulator, which provides a biphasic pulse. This protocol was developed in accordance with the guidelines for the safe use of rTMS.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham group (Sham Comparator): Sham stimulation will be performed for five consecutive days for 2 weeks (using 90% of the resting motor threshold/total of 500 pulses). For the sham stimulation a sham coil will be used.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive and painless brain stimulation technique that allows the brain excitability to change based on Faraday's Law of Electromagnetic induction . Since the presentation of the CNP is usually bilateral, the coil will be targeting the dominant hand abductor pollicis brevis (APB) muscle. If the pain is more intense in one of the arms, that arm will be targeted. This protocol was developed in accordance with the guidelines for the safe use of rTMS.

SUMMARY:
Around 80% of people with spinal cord injury (SCI) develop chronic neuropathic pain (CNP). This is a debilitating condition with major negative impacts on people's quality of life. Many treatment options have been offered (invasive stimulation, drugs) but provide limited effects and many secondary effects. There is a critical need to develop a new generation of therapies. Transcranial magnetic stimulation (TMS) is a non-invasive and painless brain stimulation technique that allows researchers to explore and change brain excitability that has shown promising effects in neuropathic pain. However there is not enough evidence of what are the long lasting effects of the different protocols. In this study, 30 SCI subjects with CNP in their hands will participate in the study. The objective is to evaluate the efficacy of real versus sham repetitive transcranial magnetic stimulation (rTMS) and investigate 1) short and long term effects on pain and 2) the behavioral and neurophysiological qualities of responders and non-responders to this treatment.This will be a randomized sham controlled trial with two groups: real or sham high frequency repetitive TMS protocol (20Hz). The protocol will be done daily for two weeks. Clinical, functional and neurophysiological evaluations will be assessed at baseline, post intervention and at 6-week follow up.

ELIGIBILITY:
Inclusion criteria:

* presence of chronic neuropathic pain at or below SCI level for at least 6 months following trauma or disease of the spinal cord.
* cervical lesion.
* CNP in the upper extremity.
* pain intensity of at least 4 out of 10 in the numerical rating scale (NRS) in the NPS both screening (baseline) and randomization (pre-evaluation).both screening (baseline) and randomization (pre-evaluation).
* stable pharmacological treatment for at least 2 weeks prior to the study and throughout the trial.
* complete or incomplete lesion.

Exclusion criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Scale (NPS) | 6 weeks
  This scale was developed to assess both the quantitative and qualitative qualities of NP. It includes 11 items, assessing global pain intensity, unpleasantness, and one item which allows the patient to describe the temporal aspects of their pain and its qualities in their own words. The remaining 8 items assess specific NP qualities: "Sharp," "Hot," "Dull," "Cold," "Sensitive," "Itchy," "Deep," and "Surface." This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Total scale from 0-10, with higher score indicating more pain.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | 6 weeks
  NRS to measure pain sensation, total score from 0-10, higher score indicates more intense pain.
Short-Form McGill Pain Questionnaire. (SF-MPQ) | 6 weeks
  The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or, 3 = severe. The SF-MPQ can be scored in several ways: a) number of words/descriptors chosen by the patient. Total scale from 0 to 45, with higher score indicating higher the pain experienced.
Present Pain Intensity (PPI) index | 6 weeks
  In the PPI index the adjectives/descriptors are ranked according to increasing intensity so each descriptor can be assigned a higher score: 0= no pain, 1=mild, 2=discomforting, 3= distressing, 4= horrible, 5= excruciating. Full range from 0 to 75, with higher score indicating higher intensity pain experienced.
Visual Analogue Scale (VAS) | 6 weeks
  The Visual Analogue Scale is the pain rating scale. Full scale from 0 to 10, with higher score indicating more pain.
The American Spinal Injury Association Impairment Scale (ASIA scale) | 6 weeks
  Upper extremity motor score (UEMS) will test the clinical motor strength from 0 to 5 of each key muscle using the ASIA scale in both arms. This sum score will range from 0 (paralyzed) to 25 (normal) in each limb (total of 50 bilaterally). Higher score indicates better health outcomes
Spinal cord independence measure (SCIM III) | 6 weeks
  Spinal cord independence measure (SCIM III) measures the ability of patients with SCI to perform everyday tasks. SCIM is used for quantitative functional outcome assessment following interventions designed to promote recovery from spinal cord injury and to increase functional achievement; it covers 19 tasks in 16 categories, with a total score range 0-100; all activities of daily living, grouped into four areas of function (subscales): Self-Care (scored 0-20), Respiration and Sphincter Management (0-40), Mobility in Room and Toilet (0-10), and Mobility Indoors and Outdoors (0-30). Higher score indicates better health outcomes.
Modified Ashworth Scale (MAS) | 6 weeks
  Modified Ashworth Scale (MAS) will measure changes in spasticity in the upper limbs after the stimulation period. For each upper limb, full Score range from 0 to 4, where lower. scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.
Beck Depression Inventory (BDI) | 6 weeks
  This questionnaire is a 21-item, selfreport rating inventory that measures characteristic attitudes and symptoms of depression. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms.
Patient's Global Impression of Change (PGIC) | 6 weeks
  Full scale from 0-7, higher score indicates better health outcomes. he patients will answer the following question: "Since beginning treatment at this program, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life related to your condition?"
Resting Motor Threshold (RMT) | 6 weeks
  Using transcranial magnetic stimulation (TMS) and electromyography (EMG) to measure RMT. Motor threshold is considered to reflect membrane-related intrinsic neuronal excitability.
Recruitment curve (RC) | 6 weeks
  Using transcranial magnetic stimulation (TMS) and electromyography (EMG) to measure RC. The median amplitude at a given intensity is thought to represent trans-synaptic excitability of the corticospinal pathways.
Short intracortical inhibition (SICI) | 6 weeks
  Using transcranial magnetic stimulation (TMS) and electromyography (EMG) to measure SICI. A single pulse TMS stimulus can be inhibited if preceded by a subthreshold conditioning stimulus 3 milliseconds apart. The SICI determines if changes in corticospinal output are related to altered intracortical excitability.
Silent period (SP): | 6 weeks
  Using transcranial magnetic stimulation (TMS) and electromyography (EMG) to measure SP. During muscle contraction, the MEP is followed by a period of silent EMG activity. Changes in intracortical inhibition are reflected in altered SP duration.
Sensory threshold (ST): | 6 weeks
  Using a constant current electrical stimulator (Digitimer), sensory threshold can be quantified. It is defined as the weakest stimulus that can be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Mar Cortes, M.D., Principal Investigator — Icahn School of Medicine
Locations (1):
- Abilities Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. For individual participant data meta-analysis. Proposals should be directed to mar.cortes@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be tbd).